CLINICAL TRIAL: NCT05595122
Title: EUS-guided Choledochoduodenostomy for Primary Drainage of Malignant Distal Biliary Obstruction: a Pilot Study Using FCSEMS Through LAMS
Brief Title: EUS-guided Choledochoduodenostomy for Primary Drainage of Malignant Distal Biliary Obstruction
Acronym: SCORPION-II-p
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Rogier P. Voermans, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL81840.029.22
Record Dates: First submitted 2022-10-22; First posted 2022-10-26 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Biliary Obstruction; Pancreas Neoplasm; Distal Cholangiocarcinoma
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): EUS-CDS using FCSEMS through LAMS
  Interventions: Device: EUS-CDS

INTERVENTIONS:
Device: EUS-CDS — EUS-CDS with FCSEMS through LAMS

SUMMARY:
A prospective single-centre pilot study investigating the feasibility and safety of EUS-guided choledochostomy as primary drainage strategy in patients with distal malignant biliary obstruction using a FCSEMS through LAMS to reduce stent dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Radiographically (CT or EUS) distal malignant bile duct obstruction
* Histology or cytology proven malignancy of the primary tumour or metastasis; onsite cytology evaluation after EUS guided fine-needle sampling that is highly suspected of a malignancy suffices
* Indication for biliary drainage; in case of a resectable tumour this should be discussed during a clinical multidisciplinary meeting
* Written informed consent

Exclusion Criteria:

* Age < 18 year
* Surgically altered anatomy after previous gastric, periampullary or duodenal resection
* Cancer extending into the antrum or proximal duodenum
* Extensive liver metastases
* WHO performance score of 4 (in bed 100% of time)
* Uncorrectable coagulopathy, defined by INR>1.5 or platelets < 50 x 10^9/L*
* Clinically relevant gastric-outlet obstruction
* Unable to complete sign informed consent

  * Inclusion is allowed after corrective treatment measures are taken, according to local protocol and treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Stentdysfunction after technical successful EUS-CDS | 6 months
  Recurrent jaundice after initial clinical success, ongoing jaundice in combination with remaining dilatation of the bile ducts, or cholangitis.

SECONDARY OUTCOMES:
Number of participants with technical success of LAMS placement | 1 day (directly after intervention)
  Successful creation of a choledochoduodenostomy using a LAMS
Number of participants with technical success of FCSEMS through LAMS | 1 day (directly after intervention)
  Successful placement of FCSEMS through LAMS.
Number of participants with clinical success | 14 days
  50% decrease or normalization of bilirubin level within 14 days of the procedure. Presumed persistant hepatic secretory failure with ongoing jaundice but decreased diameter of the bile ducts and decrease of ALT, alkaline phosphatase and gamma-glutamyl transpeptidase is not considered clinical failure of the intervention.
Procedure time | 1 day (directly after intervention)
  Is measured from introduction of endoscope in the patient until removal of endoscope after completion of the procedure. In case a fine needle aspiration (FNA) or biopsy (FNB) needs to be taken from the primary tumour to confirm malignancy, time is measured after completion of this procedure.
Adverse events | 6 months
  Are defined as any probably or definitely procedure- or admission related adverse event occurring after EUS-CDS. Severity will be recorded and graded NL81840.029.22 version 1.1 08-08-2022 SCORPION-II-pilot study 23 of 45 (mild, moderate, severe or fatal) according to the ASGE lexicon.(23) Common or expected AEs are defined according to the ASGE lexicon (including the following categories: cardiovascular, pulmonary, thromboembolic, perforation, bleeding, infection, pain).
Time to stent dysfunction | 6 months
  Is calculated from the moment of stent insertion until stent dysfunction for which a new procedure is required.
Number of re-interventions | 6 months
  Is defined as any unplanned intervention (endoscopic, intervention radiology or surgical) for an adverse event, persistent jaundice or recurrent obstructive symptoms, that is needed after EUS-CDS.
Time to start treatment (chemotherapy or surgery) | 6 months
  Is defined as the number of days after EUS-CDS until initiation of chemotherapy or surgery.
Hospitalization | 30 days
  Is defined as the number of days patient was admitted within the first 30 days after the procedure.
Survival | 6 months
  Is defined by the number of days after EUS-CDS until death. The cause of death will be registered
Costs | 6 months
  Are defined as the intramural costs that were involved with EUS-CDS, collected from the electronic hospital records and linked to the Dutch unit costs

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC location VUmc, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fritzsche JA, Fockens P, Besselink MG, Busch OR, Daams F, Wielenga MCB, Wilmink JW, Voermans RP, Van Wanrooij RLJ. Optimizing EUS-guided choledochoduodenostomy with lumen-apposing metal stents for primary drainage of malignant distal biliary obstruction (SCORPION-IIp): a prospective pilot study. Gastrointest Endosc. 2025 May;101(5):1009-1016. doi: 10.1016/j.gie.2024.10.012. Epub 2024 Oct 16. PMID 39424003